CLINICAL TRIAL: NCT00519844
Title: Assessment of Satisfaction With Growth Hormone Treatment in Children Born Small for Gestational Age: Benefits of Galenic Form of the Product
Brief Title: Growth Hormone Treatment in Children Born Small for Gestational Age: Assessment of Satisfaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHLIQUID-1670; 2005-000318-11 (EudraCT Number)
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess satisfaction with growth hormone treatment in children of both sexes born small for gestational age and who are receiving growth hormone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children treated for 3 years with Maxomat® because of small for gestational age
* Postnatal growth failure by the age of 3 years or more
* No associated growth hormone deficiency
* Height growth velocity greater than 2 cm/yr over the 12 month period preceding the inclusion
* Bone age no more than 13 years for girls and no more than 15 years for boys

Exclusion Criteria:

* Known, evolving tumour
* Hypertrophic cardiomyopathy
* Hypertension not controlled on maximum therapy
* Benign intracranial hypertension
* Known glucose intolerance or known diabetes mellitus
* Acute or active chronic hepatitis
* Chronic renal failure
* Chromosomal and/or genetic syndromes (other than Silver-Russell syndrome) or abnormality

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2005-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction/preference with the method of treatment assesses by means of a satisfaction questionnaire and a standard questionnaire of preference | after 3 months of treatment

SECONDARY OUTCOMES:
Clinical (adverse events)
Biological (fasting glucose, fasting insulin, liver enzymes)
Tolerance of the treatment
Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Lyon, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com